CLINICAL TRIAL: NCT04802733
Title: Phase 1 Study To Assess the Safety and Tolerability of Human Embryonic Stem Cell-Derived Midbrain Dopamine Neuron Cell Therapy (MSK-DA01) For Advanced Parkinson's Disease
Brief Title: Phase 1 Safety and Tolerability Study of MSK-DA01 Cell Therapy for Advanced Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BlueRock Therapeutics (Industry)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSK-DA01-101
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Advanced Parkinson's Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- MSK-DA01 (Experimental)
  Interventions: Biological: MSK-DA01; Device: MSK-DA01 Cell Delivery Device

INTERVENTIONS:
Biological: MSK-DA01 — MSK-DA01 is an experimental product derived from human embryonic stem cells. The stem cells were converted into brain cells that produce dopamine.
Device: MSK-DA01 Cell Delivery Device — A device that is used for injection of fluids into the brain will be used. Some minor modifications have been made to the device to allow delivery of MSK-DA01 cells.

SUMMARY:
This clinical trial is designed to test whether surgically injecting nerve cells that make dopamine into the brain of Parkinson's disease patients is safe, and to monitor for potential side effects.

DETAILED DESCRIPTION:
Subjects will undergo surgical transplantation of the dopamine-producing cells under general anesthesia into a part of the brain called the putamen. Subjects then take medicines to partially suppress their immune system (aimed to prevent the body from rejecting the cells) for 1 year. Safety, tolerability, evidence of cell survival (using MRI and PET scans of the brain), and effect on Parkinson's disease symptoms are assessed for 2 years post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-78 years old (Canada)
* Age 60-78 years old (United States)
* Diagnosis of Parkinson's Disease made between 3 to 20 years ago
* Taking levodopa, but with complications of therapy such as wearing off and/or dyskinesia
* Able to participate in all study visits and evaluations, including brain MRI and PET scan
* Existence of a study partner who may act as potential surrogate over long term for ongoing consent

Exclusion Criteria:

* Diagnosis of primary mitochondrial disorder, epilepsy, stroke, multiple sclerosis or other neurodegenerative diseases such as Alzheimer's disease
* Prior Deep Brain Stimulation , lesion therapy, or gene therapy for PD
* Prior surgical or radiation therapy to the brain or spinal cord
* Any medical condition resulting in high risk of immunosuppressive drugs, including any active infectious disease
* Inability to temporarily stop anti-platelet agents or other anti-coagulant medications without serious risk
* Previous or currently active malignant disease within the past 5 years, except basal cell carcinoma or in situ uterine cervical carcinoma that have been treated
* Severe obesity (>350 lbs) or any condition that prevents use of PET/MRI
* Pregnancy or breastfeeding
* Contraindication to surgery or general anesthesia
* In the opinion of the investigator, any other condition regarded as making subject unsuitable for trial

Ages: 50 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Baseline to 1 Year Post-Transplant
  The incidence of Serious Adverse Events (SAEs) at 1 year post-transplant. or abnormal tissue overgrowth related to presence of transplanted cells;

SECONDARY OUTCOMES:
Evidence of Cell Survival | Baseline to 1 Year Post-Transplant and Baseline to 2 Years Post-Transplant
  Change in 18F-DOPA uptake using positron emission tomography (PET) from baseline to 1 and 2 years
Changes in Motor Function | Baseline to 1 Year Post-Transplant and Baseline to 2 Years Post-Transplant
  Changes in MDS-Unified Parkinson's Disease Rating Scale (UPDRS) motor sub-score in the "off" state from baseline to 2 years post-transplant.
Changes in Waking Hours in "Off" State | Baseline to 1 Year Post-Transplant and Baseline to 2 Years Post-Transplant
  Changes in number of waking hours in the "off" state from baseline to 2 years post-transplant.
Continued Safety and Tolerability | Baseline to 1 Year Post-Transplant and Baseline to 2 Years Post-Transplant
  Incidence of SAEs at 2 years post-transplant and incidence and type of AEs at 1 and 2 years post-transplant.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - University of California Irvine, Orange, California
  - Weill Cornell Medical College, New York, New York
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No